CLINICAL TRIAL: NCT04270409
Title: A Phase 3 Randomized, Open-label, Multicenter Study of Isatuximab (SAR650984) in Combination With Lenalidomide and Dexamethasone Versus Lenalidomide and Dexamethasone in Patients With High-risk Smoldering Multiple Myeloma
Brief Title: Isatuximab in Combination With Lenalidomide and Dexamethasone in High-risk Smoldering Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC15992; U1111-1222-7068 (Registry Identifier: ICTRP); 2023-507419-37 (Registry Identifier: CTIS (EU)); 2019-003139-47 (EudraCT Number)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Plasma Cell Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Lenalidomide; Dexamethasone; montelukast; Acetaminophen; Diphenhydramine; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isatuximab, lenalidomide, and dexamethasone (ILd) (Experimental): Participants will receive isatuximab [intravenous (IV) administration] in combination with lenalidomide [per os (PO) administration] and dexamethasone [IV on Day 1 of Cycle 1 for participants receiving isatuximab IV only and PO otherwise for subsequent cycles] for 24 cycles followed by isatuximab monotherapy for 12 cycles for a total duration of 36 cycles. 1 cycle = 28 days. Participants may receive other treatments as pre-medication.
  Interventions: Drug: Isatuximab SAR650984; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Montelukast or equivalent; Drug: Acetaminophen; Drug: Diphenhydramine or equivalent; Drug: Methylprednisolone or equivalent
- Lenalidomide and dexamethasone (Ld) (Active Comparator): Lenalidomide [PO administration] in combination with dexamethasone [PO administration] for 24 cycles. 1 cycle = 28 days
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical for: Solution for infusion Route of administration: Intravenous
  Other Names: Sarclisa
  Arms: Isatuximab, lenalidomide, and dexamethasone (ILd)
Drug: Lenalidomide — Pharmaceutical form: Capsules Route of administration: Oral
Drug: Dexamethasone — Pharmaceutical form: Tablets and solution for injection Route of administration: Oral and intravenous
Drug: Montelukast or equivalent — Auxiliary Medicinal Product (AxMP)/pre-medication; ATC code: R03DC03; Pharmaceutical form: tablet; Route of administration: Oral;
  Arms: Isatuximab, lenalidomide, and dexamethasone (ILd)
Drug: Acetaminophen — AxMP/pre-medication ATC code: N02BE01 Pharmaceutical form: tablet/ampule/capsule; Route of administration: Intravenous (IV) or per os (PO)
  Arms: Isatuximab, lenalidomide, and dexamethasone (ILd)
Drug: Diphenhydramine or equivalent — AxMP/pre-medication ATC code: R06AA02 Pharmaceutical form: ampule; Route of administration: Intravenous
  Arms: Isatuximab, lenalidomide, and dexamethasone (ILd)
Drug: Methylprednisolone or equivalent — AxMP/pre-medication; ATC code: H02AB04; Pharmaceutical form: vial; Route of administration: Intravenous
  Arms: Isatuximab, lenalidomide, and dexamethasone (ILd)

SUMMARY:
Primary Objectives:

* Safety run-in Part: To confirm the recommended dose of isatuximab when combined with lenalidomide and dexamethasone in participants with high-risk smoldering multiple myeloma (SMM)
* Randomized Phase 3 Part: To demonstrate the clinical benefit of isatuximab in combination with lenalidomide and dexamethasone in the prolongation of progression-free survival when compared to lenalidomide and dexamethasone in subjects with high-risk SMM

Secondary Objectives:

Safety run-in Part:

* To assess overall response rate (ORR)
* To assess duration of response (DOR)
* To assess minimal residual disease (MRD) negativity in participants achieving very good partial response (VGPR) or complete response (CR)
* To assess time to diagnostic (SLiM CRAB) progression or death
* To assess time to first-line treatment for multiple myeloma (MM)
* To assess the potential immunogenicity of isatuximab
* Impact of abnormal chromosomal subtype on participant outcome

Randomized Phase 3 Part:

Key Secondary Objectives:

To compare between the arms

* MRD negativity
* Sustained MRD negativity
* Second progression-free survival (PFS2)
* Overall survival

Other Secondary Objectives:

To evaluate in both arms

* CR rate
* ORR
* DOR
* Time to diagnostic (SLiM CRAB) progression
* Time to biochemical progression
* Time to first-line treatment for MM
* Impact of abnormal chromosomal subtype on participant outcome
* Safety and tolerability
* Pharmacokinetics (PK)
* Potential of isatuximab immunogenicity
* Clinical outcome assessments (COAs)

DETAILED DESCRIPTION:
Study duration is expected to be approximately 12 years, including a 42-day screening period, followed by an up to 36-month treatment period, and a follow-up period of approximately 9 years.

ELIGIBILITY:
Inclusion criteria:

* Participants who are diagnosed within 5 years with SMM (per International Myeloma Working Group [IMWG] criteria), defined as serum M-protein ≥30 g/L or urinary M-protein ≥500 mg per 24 hour or both, and/or clonal bone marrow plasma cells (BMPCs) 10% to <60%, and absence of myeloma defining events or other related conditions and with high-risk SMM
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1 or 2
* Capable of giving voluntary written informed consent
* Absolute neutrophil count (ANC) ≥1000/µL (1 × 10^9/L)
* Platelets ≥50,000/µL (50 × 10^9/L)
* Total bilirubin ≤3 mg/dL (except Gilbert syndrome, in which direct bilirubin should be -≤5 mg/dL).
* Alanine aminotransferase ≤3× upper limit of normal (ULN), aspartate aminotransferase ≤ 3 × ULN.

Exclusion criteria:

* Evidence of any of the following calcium, renal failure, anemia, bone lesions (CRAB) criteria or Myeloma Defining Events (SLiM CRAB) detailed below (attributable to the participants SMM involvement):

  * Increased calcium levels: Corrected serum calcium >1 mg/dL above the ULN or >11 mg/dL
  * Renal insufficiency: Determined by glomerular filtration rate (GFR) <40 mL/min/1.73 m² (Modification of Diet in Renal Disease [MDRD] Formula) or serum creatinine >2 mg/dL
  * Anemia (hemoglobin 2 g/dL below lower limit of normal or <10 g/dL or both) transfusion support or concurrent treatment with erythropoietin stimulating agents is not permitted
  * ≥ 1 bone lytic lesion
  * BMPCs ≥60%
  * Serum involved/uninvolved FLC ratio ≥100 and an involved FLC ≥100mg/L
  * Whole body magnetic resonance imaging (WB-MRI) or positron emission tomography-computed tomography (PET-CT) with more than 1 bone focal lesion (≥5 mm in diameter by MRI)
* Primary systemic amyloid light-chain (AL) amyloidosis, monoclonal gammopathy of undetermined significance (MGUS), standard risk smoldering myeloma, soft tissue plasmacytoma, symptomatic myeloma
* Uncontrolled infection within 28 days prior to randomization in Phase 3 or first study intervention administration in safety run-in
* Clinically significant cardiac or vascular disease within 3 months prior to randomization, e.g. Myocardial Infarction; Unstable Angina; Coronary (e.g. Coronary Artery Bypass Graft, Percutaneous Coronary Intervention) or peripheral artery revascularization, Left Ventricular Ejection Fraction <40%, Heart Failure NYHA III-IV, Stroke, Transient Ischemic Attack, Pulmonary Embolism, other thromboembolic event, cardiac arrhythmia (Grade 3 or higher by NCI-CTCAE Version 5.0)
* Known acquired immunodeficiency syndrome (AIDS)-related illness or known human immunodeficiency virus (HIV) disease requiring antiviral treatment or active hepatitis A (defined as positive hepatitis A antigen or positive IgM). HIV serology at screening will be tested for German participants and any other country where required as per local regulations and serology hepatitis B and C at screening will be tested for all participants
* Uncontrolled or active hepatitis B virus (HBV) infection: Patients with positive Hepatitis B surface antigen (HBsAg) and/or HBV Deoxyribonucleic acid (DNA)

Of note:

* Patient can be eligible if anti-HBc Immunoglobulin G (IgG) positive (with or without positive anti-HBs) but HBsAg and HBV DNA are negative. If anti-HBV therapy in relation with prior infection was started before initiation of IMP, the anti-HBV therapy and monitoring should continue throughout the study treatment period.
* Patients with negative HBsAg and positive HBV DNA observed during screening period will be evaluated by a specialist for start of anti-viral treatment: study treatment could be proposed if HBV DNA becomes negative and all the other study criteria are still met.
* Active hepatitis C virus (HCV) infection: positive HCV ribonucleic acid (RNA) and negative anti-HCV

Of note:

* Patients with antiviral therapy for HCV started before initiation of IMP and positive HCV antibodies are eligible. The antiviral therapy for HCV should continue throughout the treatment period until seroconversion.
* Patients with positive anti-HCV and undetectable HCV RNA without antiviral therapy for HCV are eligible
* Malabsorption syndrome or any condition that can significantly impact the absorption of lenalidomide
* Any of the following within 3 months prior to randomization (or first study intervention administration in safety run-in cohort): treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism, or other uncontrolled thromboembolic event
* Received treatment (eg surgery, radiotherapy, medication) for a malignancy within 3 years of randomization (or first study intervention administration in safety run-in cohort)
* Prior exposure to approved or investigational treatments for SMM or multiple myeloma (MM) (including but not limited to conventional chemotherapies, immunomodulatory imid drugs, or Proteasome inhibitors); concurrent use of bisphosphonates or receptor activator of nuclear factor kappa-B ligand (RANKL) inhibitor denosumab is not permitted; however, prior bisphosphonates or once-a-year intravenous bisphosphonate given for the treatment of osteoporosis is permitted
* Ongoing treatment with corticosteroids with a dose >10 mg prednisone or equivalent per day at the time of randomization (or first study intervention administration in safety run-in cohort)
* Women of childbearing potential or male participant with women of childbearing potential who do not agree to use a highly effective method of birth control
* Vaccination with a live vaccine 4 weeks before the start of the study drug. Seasonal flu vaccines that do not contain live virus are permitted

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2030-10-14 (Estimated); Study Completion 2033-10-21 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent adverse events (AEs) and serious adverse events- Safety Run-in Part | Up to approximately 63 months
Plasma concentration of isatuximab during the treatment period - Safety Run-in Part | After first infusion from Cycle 1 Day 1 to Day 28 in safety run-in part
Receptor density/receptor occupancy Safety Run-in Part | Baseline to Cycle 2 Day 1 (each cycle is 28 days)
  Change in CD38 receptor occupancy from baseline
Progression-free survival (PFS) Randomized Phase 3 Part | Up to approximately 114 months
  PFS defined as the time from randomization to MM (SLiM CRAB criteria) or other related conditions based on independent review committee (IRC) assessment according to 2014 International Myeloma Working Group (IMWG) criteria or death from any cause, whichever happens first

SECONDARY OUTCOMES:
Overall Response Rate (ORR)- Safety Run-in Part | Up to approximately 63 months
  ORR defined as the proportion of participants with best overall response (BOR) recorded as partial response (PR) or better according to 2016 IMWG criteria
Duration of Response (DOR) - Safety Run-in Part | Up to approximately 63 months
  DOR defined as the time from the date of the first response to date of first progressive disease (PD) or death, whichever happens first.
Minimal residual disease (MRD) negativity -Safety Run-in Part | Up to approximately 36 months
  MRD negativity defined as the proportion of participants for whom MRD is negative in participants achieving very good partial response (VGPR) or above.
Time to diagnostic (SLiM CRAB) progression or death - Safety Run-in Part | Up to approximately 63 months
  Time to diagnostic (SLiM CRAB) progression or death defined as the time from the date of the first study intervention administration to diagnosis of SLiM CRAB or other related conditions progression or death from any cause, whichever happens first.
Time to first-line treatment for multiple myeloma (MM) - Safety Run-in Part | Up to approximately 63 months
  Time to first-line treatment for MM defined as the time from the date of the first study intervention administration to first-line treatment for MM.
Number of participants with anti-drug antibodies (ADA) against isatuximab- Safety Run-in Part | Up to approximately 63 months
PFS in participants with chromosomal abnormalities - Safety Run-In Part | Up to approximately 63 months
  Association of chromosomal abnormalities with survival outcomes
Overall Survival (OS) in participants with chromosomal abnormalities - Safety Run-In Part | Up to approximately 63 months
  Association of chromosomal abnormalities with survival outcomes
Minimal residual disease (MRD) negativity - Randomized Phase 3 Part | Up to approximately 36 months
  MRD negativity defined as the proportion Number of participants for whom MRD is negative in participants achieving VGPR or above.
Sustained MRD negativity - Randomized Phase 3 Part | Up to approximately 36 months
  Sustained MRD negativity defined as the proportion of participants for whom MRD is negative during a minimum period of one year.
Second PFS (PFS2) - Randomized Phase 3 Part | Up to approximately 144 months
  PFS2 defined as the time from the date of randomization to the date of first documentation of PD (as reported by the Investigator) after initiation of further treatment for MM or the date of death from any cause, whichever happens first
OS - Randomized Phase 3 Part | Up to approximately 114 months
  OS defined as the time from date of randomization to death from any cause.
Complete response (CR) rate - Randomized Phase 3 Part | Up to approximately 114 months
  Percentage of participants with a CR (or better [stringent CR (sCR)]) as defined by 2016 IMWG response criteria, assessed by an IRC based on central laboratory values.
Overall Response Rate (ORR) - Randomized Phase 3 Part | Up to approximately 114 months
  ORR is defined as the proportion of participants with BOR recorded as PR or better according to the 2016 IMWG criteria, assessed by an IRC based on central laboratory values.
Duration of response (DOR) - Randomized Phase 3 Part | Up to approximately 114 months
  DOR is defined as the time from the date of the first IRC determined response to the date of first IRC PD, or death, whichever happens first.
Time to diagnostic (SLiM CRAB) progression - Randomized Phase 3 Part | Up to approximately 114 months
  Time to diagnostic (SLiM CRAB) progression defined as the time from randomization to the date of diagnosis of SLiM CRAB progression based on IRC assessment.
Time to biochemical progression - Randomized Phase 3 Part | Up to approximately 114 months
  Time to biochemical progression defined as the time from randomization to the date of biochemical progression based on IRC assessment.
Time to first-line treatment for MM- Randomized Phase 3 Part | Up to approximately 144 months
  Time to first-line treatment for MM defined as the time from randomization to first-line treatment for MM
PFS in participants with chromosomal abnormalities - Randomized Phase 3 Part | Up to approximately 114 months
  Association of chromosomal abnormalities with survival outcomes.
OS in participants with chromosomal abnormalities - Randomized Phase 3 Part | Up to approximately 144 months
  Association of chromosomal abnormalities with survival outcomes.
Number of participants with Treatment-emergent adverse events (AEs) and serious adverse events - Randomized Phase 3 Part | Up to approximately 144 months
Plasma concentration of isatuximab (Ctrough)- Safety Run-in and Randomized Phase 3 Part | Baseline to Cycle 2 Day 1 (each cycle is 28 days)
  Ctrough defined as concentration observed just before treatment administration during repeated dosing after IV administration
Concentration observed at the end of intravenous infusion.(Ceoi)- Safety Run-in Part | Day 1 of Cycle 1 to 4
Number of participants with Incidence of anti-drug antibodies (ADA) against isatuximab- Randomized Phase 3 Part | Up to approximately 144 months
European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 - Randomized Phase 3 Part | Baseline to follow-up (up to approximately 114 months)
  The EORTC Multiple Myeloma Module (QLQ-C30) will be used to assess cancer-specific health related quality of life (HRQL), disease and treatment related symptoms and impact of symptoms. Mean change from baseline scores will be assessed, with responses ranging from 1=not at all to 4=very much or 1=very poor to 7=excellent; higher scores represent a better level of physical functioning
EORTC QLQ-MY20 - Randomized Phase 3 Part | Baseline to follow-up (up to approximately 114 months)
  The EORTC Multiple Myeloma Module (QLQ-MY20) will be used to measure myeloma-specific HRQL, disease and treatment related symptoms and impact of symptoms. Mean change from baseline in scores will be assessed using a 4-point scale, with responses ranging from 1=not at all to 4=very much; higher scores represent better perspectives of the future and higher level of symptomatology
EQ-5D-5L - Randomized Phase 3 Part | Baseline to follow-up (up to approximately 114 months)
  The EQ-5D-5L will be used to assess health status and health utility. Mean change from baseline scores will be assessed from 5 items, with responses ranging from 'no' to 'extreme problems'; health state utility values (HSUVs) are generated by multiplying the item scores by country specific value sets; health status is assessed via a VAS; higher scores = higher HSUV/health status
Randomized Phase 3: HRUPQ - Randomized Phase 3 Part | Baseline to follow-up (up to approximately 114 months)
  Mean change from baseline in Health resource utilization and productivity questionnaire (HRUPQ) scores. HRUPQ will assess health care resource utilization of HRSM and the impact of high risk smoldering multiple myeloma (HRSMM) on employment/work; higher scores = greater impact on work/productivity, resources.
Patient's Qualitative Assessment of Treatment Version 2 (PQAT-v2) - Randomized Phase 3 Part | End of treatment (up to approximately 3 year)
  PQAT-v2 will be used to assess participant-perceived advantages and disadvantages of treatment. Patient's qualitative assessment of treatment will be assessed using a 10 point VAS/NRS scale with response anchors of 'not beneficial at all' to 'extremely beneficial'; higher scores represent greater patient-perceived benefits of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (105):
- United States (9):
  - UCLA Site Number : 8400010, Los Angeles, California
  - Colorado Blood Cancer Institute Site Number : 8400007, Denver, Colorado
  - Cancer Specialist of North Florida Site Number : 8400011, Jacksonville, Florida
  - University of Miami Site Number : 8400012, Miami, Florida
  - Dana Farber Cancer Institute Site Number : 8400001, Boston, Massachusetts
  - Presbyterian Hospital Site Number : 8400015, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center Site Number : 8401015, Winston-Salem, North Carolina
  - Tennessee Oncology Site Number : 8400006, Nashville, Tennessee
  - ~University of Texas - MD Anderson Cancer Center Site Number : 8400002, Houston, Texas
- Australia (7):
  - Investigational Site Number :0360008, Liverpool, New South Wales
  - Investigational Site Number :0360005, Waratah, New South Wales
  - Investigational Site Number :0360001, Wollongong, New South Wales
  - Investigational Site Number :0360002, Fitzroy, Victoria
  - Investigational Site Number :0360007, Heidelberg West, Victoria
  - Investigational Site Number :0360004, Richmond, Victoria
  - Investigational Site Number :0360006, Nedlands, Western Australia
- Investigational Site Number :0760002, São Paulo, São Paulo, Brazil
- Canada (3):
  - Investigational Site Number :1240004, Edmonton, Alberta
  - Investigational Site Number :1240005, Moncton, New Brunswick
  - Investigational Site Number :1240001, Montreal, Quebec
- China (6):
  - Investigational Site Number :1560002, Hangzhou
  - Investigational Site Number :1560003, Hangzhou
  - Investigational Site Number :1560006, Nanchang
  - Investigational Site Number :1560004, Shanghai
  - Investigational Site Number :1560005, Shenyang
  - Investigational Site Number :1560001, Tianjin
- Czechia (5):
  - Investigational Site Number : 2030004, Brno
  - Investigational Site Number : 2030005, Hradec Králové
  - Investigational Site Number : 2030002, Olomouc
  - Investigational Site Number : 2030003, Ostrava - Poruba
  - Investigational Site Number : 2030001, Prague
- Denmark (4):
  - Investigational Site Number :2080001, Aalborg
  - Investigational Site Number :2080003, Aarhus N
  - Investigational Site Number :2080005, Copenhagen
  - Investigational Site Number :2080002, Roskilde
- France (9):
  - Investigational Site Number :2500009, Ars-Laquenexy
  - Investigational Site Number :2500010, Bayonne
  - Investigational Site Number :2500007, Grenoble
  - Investigational Site Number :2500006, La Roche-sur-Yon
  - Investigational Site Number :2500003, Lille
  - Investigational Site Number :2500005, Paris
  - Investigational Site Number :2500011, Paris
  - Investigational Site Number :2500002, Poitiers
  - Investigational Site Number :2500001, Rennes
- Germany (2):
  - Investigational Site Number :2760001, Hamburg
  - Investigational Site Number :2760002, Heidelberg
- Greece (3):
  - Investigational Site Number :3000002, Athens
  - Investigational Site Number :3000001, Athens
  - Investigational Site Number :3000003, Thessaloniki
- Hungary (4):
  - Investigational Site Number :3480003, Budapest
  - Investigational Site Number :3480001, Budapest
  - Investigational Site Number :3480002, Debrecen
  - Investigational Site Number :3480004, Kaposvár
- Ireland (3):
  - Investigational Site Number :3720001, Dublin, Dublin
  - Investigational Site Number :3720002, Dublin, Dublin
  - Investigational Site Number :3720003, Dublin, Dublin
- Israel (6):
  - Investigational Site Number :3760004, Ashdod
  - Investigational Site Number :3760001, Jerusalem
  - Investigational Site Number :3760002, Jerusalem
  - Investigational Site Number :3760005, Petah Tikva
  - Investigational Site Number :3760006, Ramat Gan
  - Investigational Site Number :3760003, Tel Aviv
- Italy (5):
  - Investigational Site Number :3800006, Meldola, Forlì-Cesena
  - Investigational Site Number :3800001, Rozzano, Milano
  - Investigational Site Number :3800005, Ancona
  - Investigational Site Number :3800003, Bologna
  - Investigational Site Number :3800002, Terni
- Japan (7):
  - Investigational Site Number :3920002, Nagoya, Aichi-ken
  - Investigational Site Number :3920006, Kamogawa-shi, Chiba
  - Investigational Site Number :3920008, Maebashi, Gunma
  - Investigational Site Number :3920005, Higashiibaraki-gun, Ibaraki
  - Investigational Site Number :3920003, Okayama, Okayama-ken
  - Investigational Site Number :3920009, Sunto-gun, Shizuoka
  - Investigational Site Number :3920001, Shibuya-ku, Tokyo
- Investigational Site Number :4400001, Vilnius, Lithuania
- New Zealand (2):
  - Investigational Site Number :5540004, Christchurch, Canterbury
  - Investigational Site Number :5540001, Hamilton, Waikato Region
- Norway (2):
  - Investigational Site Number :5780002, Bergen
  - Investigational Site Number :5780001, Oslo
- Poland (4):
  - Investigational Site Number :6160006, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number :6160002, Lodz, Lódzkie
  - Investigational Site Number :6160008, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number :6160005, Chorzów, Silesian Voivodeship
- South Korea (4):
  - Investigational Site Number :4100004, Gangnam-gu, Seoul-teukbyeolsi
  - Investigational Site Number :4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100002, Seoul
- Spain (7):
  - Investigational Site Number :7240004, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240006, Pamplona, Navarre
  - Investigational Site Number :7240002, Valencia, Valenciana, Comunidad
  - Investigational Site Number :7240005, Madrid
  - Investigational Site Number :7240007, Salamanca
  - Investigational Site Number :7240003, Zaragoza
- Sweden (2):
  - Investigational Site Number :7520001, Gothenburg
  - Investigational Site Number :7520003, Helsingborg
- Turkey (Türkiye) (5):
  - Investigational Site Number : 7920005, Ankara
  - Investigational Site Number : 7920001, Ankara
  - Investigational Site Number : 7920004, Istanbul
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920003, Izmir
- United Kingdom (4):
  - Investigational Site Number :8260002, Bournemouth, Hampshire
  - Investigational Site Number :8260003, London, London, City of
  - Investigational Site Number :8260001, Leicester
  - Investigational Site Number :8260004, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC15992 Plain Language Results Summaries — https://www.trialsummaries.com/Study/StudyDetails?id=25236&tenant=MT_SNY_9011